CLINICAL TRIAL: NCT00189371
Title: Reinduction Chemotherapy Containing Carboplatin and Paclitaxel With or Without Epoetin Alpha in Recurrent Platinum Sensitive Ovarian Cancer, Cancer of the Fallopian Tube or Peritoneum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.7
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Epithelial Ovarian Cancer, Fallopian Tube or Peritoneum; Platinum Sensitve Relapse; Anemia
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Anemia | interventions — Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: paclitaxel, carboplatin, epoetin alpha

SUMMARY:
Patients with epithelial ovarian cancer, fallopian tube or peritoneal cancer who receive surgical cytoreduction and platinum/taxane containing chemotherapy have a significant chance of entering complete clinical remission but about 70% will eventually relapse. Relapse more than 6 months following first line chemotherapy is regarded as platinum/taxane sensitive disease. Reinduction chemotherapy with platinum/taxane is known to be an effective treatment option. Therapy induced anemia is a common problem resulting in decrease of quality of life. The rationale of this trail is to evaluate the effects of epoetin alpha on reduction of therapy induced anemia, rate of transfusions and on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Relapse longer than 6 months after termination of platinum/taxane based first line chemotherapy
* Previously histologically confirmed cancer of: ovary, fallopian tube, peritoneum
* measurable and evaluable lesions by ultrasound, computer-tomography or MRI
* Performance status ECOG < 2 or karnofsky index > 60%
* normal organ function

Exclusion Criteria:

* more than 1 chemotherapy prior enrollment
* ongoing treatment with epoetin alpha or related drugs
* history of thrombosis or embolism during the past 12 months prior enrollment
* ileus
* left ventricular failure > NYHA classification > 2
* Ongoing toxicity of any kind (> CTC Grad II)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-02; Study Completion 2005-12

PRIMARY OUTCOMES:
Reduction of anemia

SECONDARY OUTCOMES:
Quality of life
Overall survival
Progression free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jackisch, MD, PhD, Principal Investigator — AGO Study Group
Locations (1):
- Department of Gynecology University of Marburg, Marburg, Germany

REFERENCES:
- See also: homepage of the german ovarian cancer study group AGO — http://www.ago-ovar.de